CLINICAL TRIAL: NCT04470011
Title: Survey of Procedures and Resources for Initiating Treatment of HIV in Africa: The SPRINT Study in Zambia
Brief Title: Survey of Procedures and Resources for Initiating Treatment of HIV in Africa-Zambia
Acronym: SPRINT-Zambia
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Witwatersrand, South Africa (Other); Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: H-40488; OPP1136158 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: HIV; Antiretroviral Therapy
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who initiated HIV treatment
  Interventions: Other: Routine medical record data collection
- Service providers at study facilities
  Interventions: Other: Interviews with service providers

INTERVENTIONS:
Other: Routine medical record data collection — The study will collect routine medical record data from the electronic medical record system, other electronic databases, and paper charts.
  Groups: Patients who initiated HIV treatment
Other: Interviews with service providers — Clinicians and lay staff will be interviewed regarding the ART initiation process.
  Groups: Service providers at study facilities

SUMMARY:
In its 2017 revision of the global guidelines for HIV care and treatment, the World Health Organization (WHO) called for rapid or same-day initiation of antiretroviral treatment (ART) for eligible patients testing positive for HIV. However, to date neither the WHO nor the Zambia Ministry of Health has provided detailed guidance on how to implement this recommendation.

In sub-Saharan Africa, where most HIV patients are located, studies continue to document high losses of treatment-eligible patients from care before they receive their first dose of antiretroviral medications (ARVs). Among facility-level reasons for these losses are treatment initiation protocols that require multiple clinic visits and long waiting times before a patient who tests positive for HIV is dispensed an initial supply of medications. There is very little published evidence on the practical details of the process and the extent to which it varies by facility, setting, or country. Without a robust baseline evidence base, it is challenging to identify opportunities for making improvements. The SPRINT (Survey of Procedures and Resources for Initiating Treatment of HIV in Africa) study will begin to develop this evidence base. SPRINT will combine a facility-level description of the standard of care with a retrospective record review of patients who recently initiated ART at the study sites. Data will be collected from 12 health facilities in Zambia. The survey will elicit detailed information about current procedures through structured interviews with clinic staff at the selected health facilities. The record review for a retrospective cohort of patients eligible for ART will estimate actual numbers of clinic visits, services provided, and duration of the steps for treatment initiation from start to finish. SPRINT is expected to identify differences in approaches to treatment initiation and potential opportunities for improvement.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* HIV-positive

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who became eligible for ART at a study facility between 1 July 2018 and 30 June 2019.
Sampling Method: Non-Probability Sample
Enrollment: 2189 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Average numbers of visits required to start ART | Up to 6 months after treatment eligibility determined
  Number of health system interactions required between HIV diagnosis and first dispensing of ARVs
Time to ART initiation | Up to 6 months after treatment eligibility determined
  Average number of days required between HIV diagnosis and first dispensing

SECONDARY OUTCOMES:
Proportion of patients who initiate by specified time intervals | Up to 6 months after treatment eligibility determined
  Proportion of patients who initiate ART within 0, 7, 14, and 28 days and 3 and 6 months of determination of treatment eligibility

OTHER OUTCOMES:
Procedures for ART initiation | Up to 6 months after treatment eligibility determined
  Detailed descriptive information addressing such topics as patient flow, number of required clinic visits, intervals between visits, services provided, staffing cadres involved, and record keeping systems

CONTACTS AND LOCATIONS:
Overall Officials: Sydney B Rosen, MPA, Principal Investigator — BU School of Public Health
Locations (2):
- Health Economics and Epidemiology Research Office, Johannesburg, Gauteng, South Africa
- Clinton Health Access Initiative, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huber A, Hirasen K, Brennan AT, Phiri B, Tcherini T, Mulenga L, Haimbe P, Shakwelele H, Nyirenda R, Wilson Matola B, Gunda A, Rosen S. Uptake of same-day initiation of HIV treatment in Malawi, South Africa, and Zambia as reported in routinely collected data: the SPRINT retrospective cohort study. Gates Open Res. 2023 May 2;7:42. doi: 10.12688/gatesopenres.14424.2. eCollection 2023. PMID 37153118